CLINICAL TRIAL: NCT00527319
Title: A Pilot Open Label Randomized Controlled Study to Evaluate the Dose Tolerance Safety and Efficacy of VT-122 Regimen for the Treatment of Cachexia in Subjects With Stage IV Non-Small Cell Lung Cancer
Brief Title: Regimen for the Treatment of Cachexia in Subjects With NSCLC
Acronym: VT-122
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: VT-1 CAX-001
Record Dates: First submitted 2007-08-30; First posted 2007-09-10 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2012-12

CONDITIONS: Cachexia
Keywords: NSCLC; anorexia; cachexia; grip strength; lean body mass
MeSH Terms: conditions — Cachexia; Anorexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A, control group (No Intervention): Supportive care only
- Group B, Low Dose VT-122 (Active Comparator): VT-122 (dose of etodolac: 400 mg/day) + supportive care
  Interventions: Drug: VT-122 low dose
- Group C, High Dose VT-122 (Active Comparator): VT-122 (dose of etodolac: 800 mg/day) + supportive care
  Interventions: Drug: VT-122 high dose

INTERVENTIONS:
Drug: VT-122 low dose — VT-122 low dose, dose escalated
  Arms: Group B, Low Dose VT-122
Drug: VT-122 high dose — VT-122 high dose, dose escalated
  Arms: Group C, High Dose VT-122

SUMMARY:
Cachexia is a presentation of a chronic manifestation of acute metabolic stress, a hypercatabolic nutritional state in which the normal fat and protein sparing mechanisms are not functioning and increased nutrition is not utilized.

To switch the nutritional system from a hypercatabolic to a normal nutritional state, therapy must block multi-factorial stress signaling a threshold of activation. Consistent with the synergistic hypothesis, propranolol and etodolac have been evaluated in subjects with advanced cancer demonstrating cachexia. This trial will evaluate the safety and efficacy of VT-122 in subjects with NSCLC who have hypercatabolic cachexia.

DETAILED DESCRIPTION:
The objective of this trial is to evaluate the safety and dose tolerability of VT-122 regimen and to evaluate the efficacy of VT-122 regimen

This trial is to be conducted on patients who have a diagnosis of Stage IV NSCLC, are not on chemotherapy, have lost 5% of their body weight in the previous 2 months and are deemed to be hypercatabolic.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with NSCLC
* Demonstrating average weight loss of 5% within 2 months prior to enrollment
* Heart rate of 72 bpm or greater
* Negative pregnancy test (female patients of child bearing age)
* Able to give informed consent
* Able to be administered medication
* Able to take food and defined nutritional support
* Have not been on beta-blockers for a minimum of 1 week prior to administration of the medication screening dose
* Have not undergone surgery for at least 2 weeks prior to entry into trial
* Have not been on chemotherapy, immunotherapy, biologic therapy, radio therapy, and experimental therapy for a minimum of two weeks prior to medication screening dose and during their participation in this trial
* An expected survival for a minimum of 12 weeks

Exclusion Criteria:

* Contraindication to nonsteroidal antiinflammatory drugs (NSAIDs) and beta blockers
* Blood pressure less than 100/65
* Weight loss of 15% within 2 months prior to recruitment
* Hypersensitivity reaction to the active components in VT-122
* History of myocardial infraction within the past 3 months
* Congestive heart failure (as determined by symptoms and ECG)
* A-V block of second or third degree
* Unstable angina
* Uncontrolled diabetes
* Unable to be assessed for grip strength
* A positive pregnancy test
* Chronic infection or sepsis
* History of bleeding disorders
* Patients with peripheral edema
* Patients on digoxin or other chronotropic drugs
* Patients with evidence of severe dehydration
* Patients with evidence of ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Guarino, MD, Study Director — Oxford Pharmaceutical Resources, Inc.
Locations (8):
- First Dynamic Health Care Services, Inc., Waco, Texas, United States
- India (7):
  - Rajalakshmi Nursing Home, Bangalore
  - Nizam Institute of Medical Sciences, Hyderabaad
  - Orchid Nursing Home, Kolkata
  - Shatabdi Super Specialty Hospital, Nashik
  - All India Institute of Medical Sciences, New Delhi
  - Indraprastha Apollo Hospital, New Delhi
  - Deenanath Mangeshkar Hospital, Pune

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient visit: March 23, 2007 Last patient visit: December 10, 2008
Groups:
- Group B, Low Dose VT-122: VT-122 low dose Supportive care
- Group C, High Dose VT-122: VT-122 high dose Supportive care
Period: Overall Study
Arm/Group | Group A, Control Group | Group B, Low Dose VT-122 | Group C, High Dose VT-122
Started | 12 | 12 | 13
Completed | 6 | 8 | 7
Not Completed | 6 | 4 | 6
Not completed — Withdrawal by Subject | 5 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Death | 0 | 3 | 1
Not completed — Intercurrent Medical Illness | 0 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A, Control Group | Group B, Low Dose VT-122 | Group C, High Dose VT-122 | Total
Number analyzed (Participants) | 12 | 12 | 13 | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 54.1 (12.0) | 55.1 (7.6) | 57.6 (10.4) | 55.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 3 | 12
  Male | 9 | 6 | 10 | 25
Region of Enrollment [Number; unit: participants]
  India | 12 | 12 | 13 | 37

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With a Positive Change From Baseline to Week 4 in Lean Body Mass
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Group A, Control Group | Group B, Low Dose VT-122 | Group C, High Dose VT-122
Number analyzed (Participants) | 12 | 12 | 13
participants
  <=0% | 8 | 6 | 5
  >0% to <5% | 3 | 3 | 3
  >=5% | 1 | 3 | 4
  Data Missing | 0 | 0 | 1

2. Primary Outcome: Proportion of Subjects With a Positive Change From Baseline to Week 4 in Grip Strength
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Group A, Control Group | Group B, Low Dose VT-122 | Group C, High Dose VT-122
Number analyzed (Participants) | 12 | 12 | 13
participants
  <=0% | 4 (4.03) | 8 (3.56) | 7 (6.25)
  >0% to <5% | 3 | 1 | 2
  >=5% | 5 | 3 | 4

ADVERSE EVENTS:
Arm/Group | Group A, Control Group | Group B, Low Dose VT-122 | Group C, High Dose VT-122
Serious Adverse Events (participants affected / at risk) | 0/12 | 4/12 | 3/13
Other Adverse Events (participants affected / at risk) | 7/12 | 9/12 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A, Control Group (N=12) | Group B, Low Dose VT-122 (N=12) | Group C, High Dose VT-122 (N=13)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiorespiratory Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A, Control Group (N=12) | Group B, Low Dose VT-122 (N=12) | Group C, High Dose VT-122 (N=13)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 2 (2) | 0 (0)
Crepitations (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheal Deviation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (SGPT) (Investigations) | 0 (0) | 2 (2) | 0 (0)
Aspartate Aminotransferase Increased (SGOT) (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Breath Sounds Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart Rate Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver Palpable Subcostal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less